CLINICAL TRIAL: NCT01094548
Title: A Randomized, Open-label, Phase II Study With Stimuvax® (L-BLP25 or BLP25 Liposome Vaccine) in Subjects With Either Chemotherapy-naïve, Slowly Progressive, Asymptomatic Multiple Myeloma or With Stage II/III Multiple Myeloma in Stable Response/Plateau Phase Following Anti-tumor Therapy
Brief Title: Study of Tecemotide (L-BLP25) in Subjects With Slowly Progressive Multiple Myeloma With no Symptoms and Who Have Had no Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR63325-008
Record Dates: First submitted 2010-03-24; First posted 2010-03-29 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-01

CONDITIONS: Multiple Myeloma
Keywords: L-BLP25 liposome; Multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — L-BLP25; Single Person; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tecemotide (L-BLP25) plus single low dose cyclophosphamide (Experimental)
  Interventions: Biological: Tecemotide (L-BLP25); Drug: Single low dose cyclophosphamide
- Tecemotide (L-BLP25) plus multiple low dose cyclophosphamide (Experimental)
  Interventions: Biological: Tecemotide (L-BLP25); Drug: Multiple low dose cyclophosphamide

INTERVENTIONS:
Biological: Tecemotide (L-BLP25) — After receiving single low dose of cyclophosphamide, subjects will receive 8 consecutive weekly subcutaneous vaccinations with 806 microgram (mcg) of tecemotide (L-BLP25) at Weeks 1, 2, 3, 4, 5, 6, 7 and 8 followed by maintenance vaccinations (806 mcg of tecemotide (L-BLP25) at 6-Week intervals, commencing at Week 14, until disease progression requiring anti-tumor therapy is documented.
  Other Names: Stimuvax
  Arms: Tecemotide (L-BLP25) plus single low dose cyclophosphamide
Biological: Tecemotide (L-BLP25) — After receiving multiple low dose of cyclophosphamide, subjects will receive 8 consecutive weekly subcutaneous vaccinations with 806 mcg of tecemotide (L-BLP25) at Weeks 1, 2, 3, 4, 5, 6, 7 and 8 followed by maintenance vaccinations (806 mcg of tecemotide (L-BLP25) at 6-Week intervals, commencing at Week 14, until disease progression requiring anti-tumor therapy is documented.
  Other Names: Stimuvax
  Arms: Tecemotide (L-BLP25) plus multiple low dose cyclophosphamide
Drug: Single low dose cyclophosphamide — An intravenous (IV) infusion of 300 milligram per square meter (mg/m^2) (to a maximum 600 mg) of cyclophosphamide will be given 3 days before the first vaccine treatment.
  Arms: Tecemotide (L-BLP25) plus single low dose cyclophosphamide
Drug: Multiple low dose cyclophosphamide — An IV infusion of 300 mg/m^2 (to a maximum 600 mg) of cyclophosphamide will be given 3 days before the first vaccine treatment plus an intravenous dose of cyclophosphamide (300 mg/m^2, to a maximum of 600 mg) 3 days prior to the tecemotide (LBLP25) administration at week 5 of the weekly treatment phase and 3 days prior to every tecemotide (L-BLP25) administration during the treatment phase with 6-Weekly administration of tecemotide (L-BLP25), commencing at Week 14 up to a maximum treatment period of 2 years.
  Arms: Tecemotide (L-BLP25) plus multiple low dose cyclophosphamide

SUMMARY:
Tecemotide (L-BLP25) is believed to induce a Mucinous glycoprotein 1 (MUC1)-specific T-cell response after vaccination. The primary purpose of this study is to ascertain whether vaccination with tecemotide (L-BLP25) induces a MUC1-specific T-cell response in slowly progressive or chemotherapy naive multiple myeloma subjects.

ELIGIBILITY:
Inclusion Criteria:

* Documented previously untreated, Mucinous glycoprotein 1 (MUC1)-expressing, slowly progressive asymptomatic multiple myeloma with an increasing M-protein concentration displayed on two occasions separated by an interval of at least 4 weeks within the last 18 months, or
* Documented MUC1-expressing stage II or III multiple myeloma with a treatment-free interval of at least 3 months following prior anti-tumor therapy, and fulfilling criteria for having a stable response/plateau phase
* Signed written informed consent
* MUC1-expressing myeloma cells in the bone marrow
* Greater than or equal to (>=) 18 years of age
* Life expectancy of at least 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to (<=) 1 at study entry
* Effective contraception for both male and female subjects, if the possibility of conception exists
* A platelet count >=100 x 10^9/Liter, white blood cells >=2.5 x 10^9/Liter, and hemoglobin >=90 gram per liter (g/L)
* Total bilirubin <= 1.5 x upper reference range
* Aspartate aminotransferase (AST) <= 2.5 x upper reference range
* Serum creatinine <= 2 x upper reference

Exclusion Criteria:

Pre-Therapies:

* Previous exposure to MUC1 targeting therapy
* Radiotherapy or any investigational drug in the 30 days before the start of treatment in this study
* Receipt of immunotherapy (Example: interferons, tumor necrosis factor [TNF], interleukins, or biological response modifiers [granulocyte macrophage colony stimulating factor {GM-CSF}, granulocyte colony stimulating factor {G-CSF}, macrophage-colony stimulating factor {M-CSF}], monoclonal antibodies) within 4 weeks (28 days) prior to randomization
* Any preexisting medical condition requiring chronic oral or intravenous steroid or immunosuppressive therapy except for maintenance doses of prednisone of <=10 milligram per day (mg/day)

Medical Conditions:

* Autoimmune disease that in the opinion of the investigator could compromise the safety of the subject in this study
* Hereditary or congenital immunodeficiencies
* Known hypersensitivity reaction to any of the components of study treatments
* Clinically significant cardiac disease, Example: New York Heart Association (NYHA) classes III-IV; unstable angina, uncontrolled arrhythmia or uncontrolled hypertension, myocardial infarction in the previous 6 months
* Other previous malignancies within 5 years, with exception of a history of a previous basal cell carcinoma of the skin, carcinoma in situ of uterine cervix, gastrointestinal intramucosal carcinoma
* Known Hepatitis B and/or C
* Splenectomy

Standard Safety:

* Known alcohol or drug abuse
* Medical or psychological conditions that would not permit the subject to complete the study or sign informed consent
* Significant disease which, in the investigator's opinion, would exclude the subject from the study
* Pregnant or breast-feeding women, women of childbearing potential, unless using effective contraception as determined by the investigator. Subjects whom the investigator considers may be at risk of pregnancy will have a pregnancy test performed per institutional standard
* Participation in another clinical study within the past 30 days
* Legal incapacity or limited legal capacity
* Concurrent treatment with a non-permitted drug
* Any other reason that, in the opinion of the investigator, precludes the subject from participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-01; Primary Completion 2011-02 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Please Contact the Merck KGaA Communication Center, Darmstadt, Germany

REFERENCES:
- [Background] Rossmann E, Österborg A, Löfvenberg E, et al. Randomized Phase II Study of BLP25 Liposome Vaccine (L-BLP25) in Patients with Multiple Myeloma. Am Soc Hematol. 53rd Annual Meeting, Dec 2011, Poster 2927.
- [Derived] Rossmann E, Osterborg A, Lofvenberg E, Choudhury A, Forssmann U, von Heydebreck A, Schroder A, Mellstedt H. Mucin 1-specific active cancer immunotherapy with tecemotide (L-BLP25) in patients with multiple myeloma: an exploratory study. Hum Vaccin Immunother. 2014;10(11):3394-408. doi: 10.4161/hv.29918. PMID 25483677

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last participant (informed consent): 21 January 2008/11 January 2010. Last participant completed: 07 March 2012; Clinical data cut-off date: 07 March 2012.
Pre-assignment Details: A total of 36 participants were screened for eligibility; 2 were excluded (mainly non-fulfillment of inclusion or exclusion) and 34 participants were enrolled and randomized.
Groups:
- Tecemotide (L-BLP25) Plus Single Low Dose Cyclophosphamide: Tecemotide (L-BLP25): After receiving single low dose cyclophosphamide, participants received 8 consecutive weekly subcutaneous vaccinations with 806 microgram (mcg) of tecemotide (L-BLP25) at Weeks 1, 2, 3, 4, 5, 6, 7 and 8 followed by maintenance vaccinations (806 mcg of tecemotide (L-BLP25) at 6-Week intervals, commencing at Week 14, until disease progression requiring anti-tumor therapy was documented.
  Single low dose cyclophosphamide: An intravenous (IV) infusion of 300 milligram per square meter (mg/m^2) (to a maximum 600 mg) of cyclophosphamide was given 3 days before the first vaccine treatment.
- Tecemotide (L-BLP25) Plus Multiple Low Dose Cyclophosphamide: Tecemotide (L-BLP25): After receiving multiple low dose cyclophosphamide, participants received 8 consecutive weekly subcutaneous vaccinations with 806 mcg of tecemotide (L-BLP25) at Weeks 1, 2, 3, 4, 5, 6, 7 and 8 followed by maintenance vaccinations (806 mcg of tecemotide(L-BLP25) at 6-Week intervals, commencing at Week 14, until disease progression requiring anti-tumor therapy was documented.
  Multiple low dose cyclophosphamide: An IV infusion of 300 mg/m^2 (to a maximum 600 mg) of cyclophosphamide was given 3 days before the first vaccine treatment plus an IV dose of cyclophosphamide (300 mg/m^2, to a maximum of 600 mg) 3 days prior to the tecemotide(LBLP25) administration at week 5 of the weekly treatment phase and 3 days prior to every tecemotide (L-BLP25) administration during the treatment phase with 6-Weekly administration of tecemotide (L-BLP25), commencing at Week-14 up to a maximum treatment period of 2 years.
Period: Overall Study
Arm/Group | Tecemotide (L-BLP25) Plus Single Low Dose Cyclophosphamide | Tecemotide (L-BLP25) Plus Multiple Low Dose Cyclophosphamide
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all the randomized participants who received at least 1 dose of trial treatment.
Groups:
- Tecemotide (L-BLP25) Plus Single Low Dose Cyclophosphamide: Tecemotide (L-BLP25): After receiving single low dose cyclophosphamide, participants received 8 consecutive weekly subcutaneous vaccinations with 806 mcg of tecemotide (L-BLP25) at Weeks 1, 2, 3, 4, 5, 6, 7 and 8 followed by maintenance vaccinations (806 mcg of tecemotide [L-BLP25]) at 6-Week intervals, commencing at Week 14, until disease progression requiring anti-tumor therapy was documented.
  Single low dose cyclophosphamide: An intravenous (IV) infusion of 300 milligram per square meter (mg/m^2) (to a maximum 600 mg) of cyclophosphamide was given 3 days before the first vaccine treatment.
- Tecemotide (L-BLP25) Plus Multiple Low Dose Cyclophosphamide: Tecemotide (L-BLP25): After receiving multiple low dose cyclophosphamide, participants received 8 consecutive weekly subcutaneous vaccinations with 806 mcg of tecemotide (L-BLP25) at Weeks 1, 2, 3, 4, 5, 6, 7 and 8 followed by maintenance vaccinations (806 mcg of tecemotide [L-BLP25]) at 6-Week intervals, commencing at Week 14, until disease progression requiring anti-tumor therapy was documented.
  Multiple low dose cyclophosphamide: An IV infusion of 300 mg/m^2 (to a maximum 600 mg) of cyclophosphamide was given 3 days before the first vaccine treatment plus an IV dose of cyclophosphamide (300 mg/m^2, to a maximum of 600 mg) 3 days prior to the tecemotide(LBLP25) administration at week 5 of the weekly treatment phase and 3 days prior to every tecemotide (L-BLP25) administration during the treatment phase with 6-Weekly administration of tecemotide (L-BLP25), commencing at Week-14 up to a maximum treatment period of 2 years.
- Total: Total of all reporting groups
Arm/Group | Tecemotide (L-BLP25) Plus Single Low Dose Cyclophosphamide | Tecemotide (L-BLP25) Plus Multiple Low Dose Cyclophosphamide | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (7.26) | 63.9 (9.36) | 63.2 (8.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Induced Mucinous Glycoprotein-1 (MUC-1)-Specific Immune Response
Description: The overall immune response was achieved at least for 2 timepoints; that is at least 1 parameter in at least 1 assay (Lymphoproliferation assay, enzyme-linked immunospot (ELISPOT) for interferon [IFN] gamma, and intracellular IFN gamma cytokine assay in peripheral blood mononuclear cell [PBMC]) with ratio to background >=2, and ratio of background-corrected value to baseline >=2;Specific immune response at a given timepoint 't' was considered as differences of log-scale values under stimulation (X vax,t ) to those of the respective unstimulated controls (Xneg,t, background values)were computed after certain assay-specific pre-processing steps: Yt = Xvax,t - Xneg,t; A participant was considered to show positive stimulation-induced immune response at timepoint 't' (POS[t]=1), upon fulfilling the following criteria: Yt =>1 (That is at least a 2-fold higher value under stimulation than without stimulation). AVvax,t-1SEM vax,t > AVneg,t+1SEMneg,t (ELISPOT and proliferation assay only).
Time Frame: From the date of randomization up to Week 104
Population: Immunological diagnostic analysis set was defined as the subset of safety analysis set consisting of all the participants with at least one complete set of baseline (baseline/cyclophosphamide infusion visit or both), Week 5, and Week 9 data of either ELISPOT, proliferation assay or cytokine assay.
Measure: Number; unit: participants
Groups:
- Tecemotide (L-BLP25) Plus Multiple Low Dose Cyclophosphamide: Tecemotide (L-BLP25): After receiving multiple low dose cyclophosphamide, participants received 8 consecutive weekly subcutaneous vaccinations with 806 mcg of tecemotide (L-BLP25) at Weeks 1, 2, 3, 4, 5, 6, 7 and 8 followed by maintenance vaccinations (806 mcg of tecemotide(L-BLP25) at 6-Week intervals, commencing at Week 14, until disease progression requiring anti-tumor therapy was documented.
  Multiple low dose cyclophosphamide: An IV infusion of 300 mg/m^2 (to a maximum 600 mg) of cyclophosphamide was given 3 days before the first vaccine treatment plus an IV dose of cyclophosphamide (300 mg/m^2, to a maximum of 600 mg) 3 days prior to the tecemotide(LBLP25) administration in Weeks 1 and 5 of the weekly treatment phase and 3 days prior to every tecemotide (L-BLP25) administration during the treatment phase with 6-Weekly administration of tecemotide (L-BLP25), commencing at Week-14 up to a maximum treatment period of 2 years.
Arm/Group | Tecemotide (L-BLP25) Plus Single Low Dose Cyclophosphamide | Tecemotide (L-BLP25) Plus Multiple Low Dose Cyclophosphamide
Number analyzed (Participants) | 17 | 15
participants | 8 | 7
Statistical Analysis 1: Comparison: Tecemotide (L-BLP25) Plus Single Low Dose Cyclophosphamide vs Tecemotide (L-BLP25) Plus Multiple Low Dose Cyclophosphamide; Test type: Superiority or Other; p = 1.0000, Fisher Exact

2. Secondary Outcome: Number of Participants With Baseline Immune Response and Initial Increase of MUC1 Specific Immune Response
Description: Baseline immune response towards MUC1 was defined as an immune response towards BP25, MUC-A2 or MUC-A11 peptide stimulation which was present in at least one of the two baseline assessments; the specific immune responses at baseline were based on the averaged baseline values across the two baseline visits. Initial increase of MUC1-specific immune response was defined as an increase of MUC1-specific immune response during the primary treatment period (up to Week 9).
Time Frame: Baseline and Week 9
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- Tecemotide (L-BLP25) Plus Multiple Low Dose Cyclophosphamide: Tecemotide (L-BLP25): After receiving multiple low dose cyclophosphamide, participants received 8 consecutive weekly subcutaneous vaccinations with 806 mcg of tecemotide (L-BLP25) at Weeks 1, 2, 3, 4, 5, 6, 7 and 8 followed by maintenance vaccinations (806 mcg of tecemotide(L-BLP25) at 6-Week intervals, commencing at Week 14, until disease progression requiring anti-tumor therapy was documented.
  Multiple low dose cyclophosphamide: An IV infusion of 300 mg/m^2 (to a maximum 600 mg/m^2) of cyclophosphamide was given 3 days before the first vaccine treatment plus an IV dose of cyclophosphamide (300 mg/m^2, to a maximum of 600 mg) 3 days prior to the tecemotide(LBLP25) administration at week 5 of the weekly treatment phase and 3 days prior to every tecemotide (L-BLP25) administration during the treatment phase with 6-Weekly administration of tecemotide (L-BLP25), commencing at Week-14 up to a maximum treatment period of 2 years.
Arm/Group | Tecemotide (L-BLP25) Plus Single Low Dose Cyclophosphamide | Tecemotide (L-BLP25) Plus Multiple Low Dose Cyclophosphamide
Number analyzed (Participants) | 17 | 15
participants
  Baseline immune response | 10 | 7
  MUC1 specific immune response at Week 9 | 8 | 7

3. Secondary Outcome: Number of Participants With Overall Induced Immune Response by Human Leukocyte-associated Antigen (HLA) Type
Description: Relationship between immune response with HLA subtypes was determined by analyzing the number of participants with overall induced immune response grouped by the presence versus absence of the given HLA type.
Time Frame: From the date of randomization up to Week 104
Population: Immunological diagnostic analysis set was defined as the subset of safety analysis set consisting of all the participants with at least 1 complete set of baseline, Week 5, and Week 9 data of either ELISPOT, proliferation assay or cytokine assay. "n" signifies number of participants evaluable for the particular HLA type, respectively.
Measure: Number; unit: participants
Arm/Group | Tecemotide (L-BLP25) Plus Single Low Dose Cyclophosphamide | Tecemotide (L-BLP25) Plus Multiple Low Dose Cyclophosphamide
Number analyzed (Participants) | 17 | 15
participants
  HLA A01 (n=3, 7) | 2 | 3
  HLA A01 not present (n=14, 8) | 6 | 4
  HLA A02 present (n=10, 10) | 5 | 4
  HLA A02 not present (n=7, 5) | 3 | 3
  HLA A03 present (n=4, 3) | 3 | 0
  HLA A03 not present (n=13, 12) | 5 | 7
  HLA A24 present (n=7, 1) | 3 | 1
  HLA A24 not present (n=10, 14) | 5 | 6
  HLA A68 present (n=2, 3) | 0 | 2
  HLA A68 not present (n=15, 12) | 8 | 5
  HLA B07 present (n=6, 5) | 3 | 2
  HLA B07 not present (n=11, 10) | 5 | 5
  HLA B08 present (n=3, 6) | 2 | 3
  HLA B08 not present (n=14, 9) | 6 | 4
  HLA B15 present (n=4, 1) | 1 | 0
  HLA B15 not present (n=13, 14) | 7 | 7
  HLA B27 present (n=3, 2) | 1 | 1
  HLA B27 not present (n=14, 13) | 7 | 6
  HLA B35 present (n=2, 4) | 2 | 2
  HLA B35 not present (n=15, 11) | 6 | 5
  HLA B44 present (n=4, 2) | 2 | 2
  HLA B44 not present (n=13, 13) | 6 | 5
  HLA C01 present (n=1, 4) | 1 | 3
  HLA C01 not present (n=16, 11) | 7 | 4
  HLA C02 present (n=3, 1) | 1 | 0
  HLA C02 not present (n=14, 14) | 7 | 7
  HLA C03 present (n=9, 2) | 4 | 0
  HLA C03 not present (n=8, 13) | 4 | 7
  HLA C04 present (n=1, 3) | 1 | 2
  HLA C04 not present (n=16, 12) | 7 | 5
  HLA C07 present (n=12, 10) | 6 | 4
  HLA C07 not present (n=5, 5) | 2 | 3
  HLA DQB02 present (n=2, 6) | 0 | 3
  HLA DQB02 not present (n=15, 9) | 8 | 4
  HLA DQB03 present (n=11, 9) | 6 | 5
  HLA DQB03 not present (n=6, 6) | 2 | 2
  HLA DQB05 present (n=6, 2) | 2 | 0
  HLA DQB05 not present (n=11, 13) | 6 | 7
  HLA DQB06 present (n=7, 5) | 4 | 3
  HLA DQB06 not present (n=10, 10) | 4 | 4
  HLA DRB01 present (n=3, 1) | 1 | 0
  HLA DRB01 not present (n=14, 14) | 7 | 7
  HLA DRB03 present (n=2, 6) | 0 | 3
  HLA DRB03 not present (n=15, 9) | 8 | 4
  HLA DRB04 present (n=11, 6) | 6 | 3
  HLA DRB04 not present (n=6, 9) | 2 | 4
  HLA DRB11 present (n=2, 5) | 1 | 3
  HLA DRB11 not present (n=15, 10) | 7 | 4
  HLA DRB13 present (n=5, 2) | 3 | 1
  HLA DRB13 not present (n=12, 13) | 5 | 6
  HLA DRB15 present (n=5, 3) | 3 | 2
  HLA DRB15 not present (n=12, 12) | 5 | 5

4. Secondary Outcome: Percentage of Participants With Objective Clinical Response (Complete Response [CR], or Partial Response [PR], or Minimal Response [MR]
Description: OCR (CR, or PR, or MR or NC or PD or NE) was defined per Blade Criteria. OCR rate (CR, or PR, or MR) was defined as the number of participants having experienced at least once a CR, PR, or MR, divided by the number of all participants. CR: negative immunofixation on serum and urine monoclonal paraprotein (M-protein), disappearance of any soft tissue plasmacytomas (STP), <=5% plasma cells in bone marrow (BM); PR: >=50% reduction in serum M-protein, plasma cells in BM, size of STP; >=90% reduction of urinary M-protein in 24 hours, no increase in size/number of the lytic bone lesions (LBL). MR: 25%-49% reduction in serum M-protein, plasma cells in BM aspirate in non-secretory myeloma participants, size of STP; 50%-89% reduction in 24 h urinary light chain reaction (LCR), and no increase in size/number of LBL. PD: >25% increase in the serum M-protein level, 24 hour urinary LCR. Increase in size of existing BL or STP, development of new BL or STP, or development of hypercalcemia
Time Frame: From the date of randomization up to Month 48
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Tecemotide (L-BLP25) Plus Single Low Dose Cyclophosphamide | Tecemotide (L-BLP25) Plus Multiple Low Dose Cyclophosphamide
Number analyzed (Participants) | 17 | 15
Percentage of participants
  CR+PR+MR | 0.0 | 0.0
  CR | 0.0 | 0.0
  PR | 0.0 | 0.0
  MR | 0.0 | 0.0

5. Secondary Outcome: Time to Progression (TTP)
Description: Progression was defined as follows per Blade criteria: The disease was considered to be progressive if it met 1 or more of the following: >25% increase in the level of serum monoclonal paraprotein (M-protein);>25% increase in the 24 h urinary light chain excretion; >25% increase in plasma cells in the bone marrow- definite increase in the size of existing bone lesions or soft tissues plasmacytomas (STP); Development of new bone lesions or STP, or development of hypercalcemia. TTP was defined as time from randomization to disease progression. Participants without events were censored on the date of last tumor assessment. Participants without PD at time of treatment discontinuation were censored at the date of discontinuation. Participants without PD at the time of the analysis but still on treatment were censored at the date of the latest available multiple myeloma status assessment. Participants dying from causes other than PD were treated as censored observations at time of death.
Time Frame: From the date of randomization up to Month 48
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tecemotide (L-BLP25) Plus Single Low Dose Cyclophosphamide | Tecemotide (L-BLP25) Plus Multiple Low Dose Cyclophosphamide
Number analyzed (Participants) | 17 | 15
months | 15.2 [14.5 to 20.8] | 38.9 [17.3 to NA] — The number of events were not sufficient to calculate the upper limit of the confidence interval.
Statistical Analysis 1: Comparison: Tecemotide (L-BLP25) Plus Single Low Dose Cyclophosphamide vs Tecemotide (L-BLP25) Plus Multiple Low Dose Cyclophosphamide; Test type: Superiority or Other; p = 0.0940, Log Rank; Hazard Ratio (HR) = 0.431, 95% CI 2-sided [0.157 to 1.185]

6. Secondary Outcome: Time to Anti-tumor Therapy
Description: Time from date of randomization to the date of first anti-tumor therapy since end of study treatment. In case a concomitant or concurrent procedure was identified as anti-tumor therapy during the medical review process, the start date of that anti-tumor therapy was used instead. Participants in the survival follow-up phase without subsequent anti-tumor therapy at the time of the analysis were censored at the latest available follow-up date. Participants without anti-tumor therapy and still on treatment at the time of analysis were censored at the data cut-off date if any trial treatment administration was recorded after the data cut-off date. In case no such record exists, the subject was censored at the last available administration date prior or equal to the data cut-off date. Participants dying before start of subsequent anti-tumor therapy were treated as censored observations at time of death.
Time Frame: From the date of randomization up to Month 48
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tecemotide (L-BLP25) Plus Single Low Dose Cyclophosphamide | Tecemotide (L-BLP25) Plus Multiple Low Dose Cyclophosphamide
Number analyzed (Participants) | 17 | 15
months | 24.7 [14.8 to NA] — The number of events were not sufficient to calculate the upper limit of the confidence interval. | 36.7 [23.3 to NA] — The number of events were not sufficient to calculate the upper limit of the confidence interval.
Statistical Analysis 1: Comparison: Tecemotide (L-BLP25) Plus Single Low Dose Cyclophosphamide vs Tecemotide (L-BLP25) Plus Multiple Low Dose Cyclophosphamide; Test type: Superiority or Other; p = 0.3919, Log Rank; Hazard Ratio (HR) = 0.666, 95% CI 2-sided [0.261 to 1.698]

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs),Serious TEAEs, TEAEs of Grade 3 or 4 According to NCI-CTCAE v3.0, TEAEs Leading to Discontinuation and Injection Site Reactions (ISRs)
Description: TEAEs occurred between the first dose of study drug administration and up to 42 days after the last dose of study drug administration that were absent before treatment or that worsened relative to pretreatment state. A Serious TEAE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect.Grade 3 and 4 TEAES as per National Cancer Institute Common Terminology Criteria for Adverse Experience version 3 (NCI-CTCAE v3.0) were presented. Grade 3 refers to severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care and Activity of daily living (ADL).Grade 4 refers to Life-threatening consequences; where urgent intervention indicated. Injection site reactions, term used per NCI-CTCAE, were also presented.
Time Frame: From the first dose of study drug administration up to 42 days after the last dose of study drug administration or clinical data cut-off date (07 March 2012)
Population: Safety analysis set included all the randomized participants who received at least 1 dose of trial treatment.
Measure: Number; unit: participants
Arm/Group | Tecemotide (L-BLP25) Plus Single Low Dose Cyclophosphamide | Tecemotide (L-BLP25) Plus Multiple Low Dose Cyclophosphamide
Number analyzed (Participants) | 17 | 17
participants
  TEAEs | 17 | 17
  Serious TEAEs | 6 | 5
  NCI-CTC Grade 3 and 4 TEAEs | 5 | 8
  TEAEs leading to discontinuation of treatment | 1 | 2
  ISRs | 8 | 11

ADVERSE EVENTS:
Time Frame: From the first dose of study drug and up to 42 days after the last dose of study drug or clinical data cut-off date (07 March 2012)
Arm/Group | Tecemotide (L-BLP25) Plus Single Low Dose Cyclophosphamide | Tecemotide (L-BLP25) Plus Multiple Low Dose Cyclophosphamide
Serious Adverse Events (participants affected / at risk) | 6/17 | 5/17
Other Adverse Events (participants affected / at risk) | 17/17 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tecemotide (L-BLP25) Plus Single Low Dose Cyclophosphamide (N=17) | Tecemotide (L-BLP25) Plus Multiple Low Dose Cyclophosphamide (N=17)
Atrial fibrillation (Cardiac disorders) | 0 | 2
Retinal detachment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 2
Wound infection (Infections and infestations) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Encephalitis (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Status epilepticus (Nervous system disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tecemotide (L-BLP25) Plus Single Low Dose Cyclophosphamide (N=17) | Tecemotide (L-BLP25) Plus Multiple Low Dose Cyclophosphamide (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 3
Dacryostenosis acquired (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 2 | 8
Diarrhoea (Gastrointestinal disorders) | 2 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gingivitis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 12
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1
Tongue blistering (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 1 | 1
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 3 | 4
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 9 | 11
Influenza like illness (General disorders) | 0 | 2
Injection site erythema (General disorders) | 3 | 4
Injection site nodule (General disorders) | 5 | 7
Injection site pruritus (General disorders) | 3 | 0
Injection site rash (General disorders) | 1 | 0
Injection site ulcer (General disorders) | 1 | 0
Injection site warmth (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 4
Allergy to arthropod bite (Immune system disorders) | 2 | 0
Seasonal allergy (Immune system disorders) | 1 | 0
Borrelia infection (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0
Eczema infected (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 1 | 1
Gastric infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 2
Gastrointestinal infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Herpes zoster ophthalmic (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Injection site abscess (Infections and infestations) | 1 | 0
Injection site infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 7 | 7
Otitis externa (Infections and infestations) | 2 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Respiratory moniliasis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 10
Urinary tract infection (Infections and infestations) | 2 | 0
Viral infection (Infections and infestations) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Back injury (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 1
Wrong drug administered (Injury, poisoning and procedural complications) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Appetite disorder (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 5
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1
Formication (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 3
Hypoaesthesia (Nervous system disorders) | 1 | 1
Migraine with aura (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 4 | 2
Insomnia (Psychiatric disorders) | 2 | 3
Mood altered (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1
Albuminuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Breast mass (Reproductive system and breast disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 3
Blood blister (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 4
Skin nodule (Skin and subcutaneous tissue disorders) | 1 | 2
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 4
Hypotension (Vascular disorders) | 0 | 1
Ectropion (Eye disorders) | 0 | 1
Injection site haematoma (General disorders) | 1 | 4
Skin bacterial infection (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Eye injury (Injury, poisoning and procedural complications) | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 0 | 1
Tumor invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bipolar disorder (Psychiatric disorders) | 0 | 1
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publications of the results, either in part or in total (abstracts in journals or newspapers, oral presentations, etc.) by Investigators or their representatives will require pre-submission review by the Sponsor. The Sponsor is entitled to delay publication in order to obtain patent protection.